CLINICAL TRIAL: NCT03605927
Title: CD40-L Blockade for Prevention of Acute Graft-Versus-Host Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCC-19305
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Graft-versus-host-disease; GVHD; GVHD, Acute
Keywords: HCT; hematopoietic cell transplantation; antibody therapy
MeSH Terms: conditions — Graft vs Host Disease | interventions — Sirolimus; Standard of Care; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Therapy (Experimental): BMS-986004: From day 13, intravenously (IV) every 2 week through day 100 post HCT.
  Tacrolimus: From day -3 as standard of care. Sirolimus: From day -1 as standard of care.
  Interventions: Drug: BMS-986004; Drug: Sirolimus; Drug: Tacrolimus

INTERVENTIONS:
Drug: BMS-986004 — BMS-986004 will be administered in ascending dose cohorts in the phase I component of the trial. Based on prior PK and PD data, dose levels of 225 mg, 675 mg, and 1500 mg (3 total phase I dose levels) will be examined. BMS-986004 will be given intravenously (IV) every 2 weeks, starting from day -3 (i.e., three days prior to HCT) onward through a total of 100 days post-HCT. The maximum tolerated dose (MTD) identified in the phase I component of the trial will be carried forward as the recommended dose level in the phase 1 expansion cohort.
  Other Names: Anti-CD40L Domain Antibody
Drug: Sirolimus — Sirolimus and tacrolimus (standard of care pharmacologic immune suppression) will be given according to institutional standards.
  Sirolimus (SIR) will be given as a loading dose on day -1 orally, then daily as maintenance therapy with target levels of 10-14ng/mL early post-HCT, then tapered to 5-14ng/mL range.
  Program standards will be used for SIR and TAC level monitoring frequency and dose adjustments, including careful attention to drug-interactions.
  Other Names: Standard of Care; SIR
Drug: Tacrolimus — Sirolimus and tacrolimus (standard of care pharmacologic immune suppression) will be given according to institutional standards.
  In brief, tacrolimus (TAC) will be started on day -3 IV, and transitioned to oral TAC when oral medications are tolerated; target level is 3-7ng/mL.
  Program standards will be used for SIR and TAC level monitoring frequency and dose adjustments, including careful attention to drug-interactions.
  Other Names: Standard of Care; TAC

SUMMARY:
The purpose of this study is to examine the safety and efficacy of the addition of BMS-986004 to standard of care Sirolimus (SIR)-based immune suppression.

DETAILED DESCRIPTION:
The approach builds upon extensive evidence supporting the benefit of CD40L blockade in disrupting key signaling events associated with immune activation. The trial addresses a pressing clinical need, namely prevention of Graft-Versus-Host Disease (GVHD) after hematopoietic cell transplantation (HCT) and promotion of donor-recipient immune tolerance. The safety profile of this anti-CD40L antibody overcomes major prior limitations, and the planned biologic studies will provide significant mechanistic insight.

ELIGIBILITY:
Inclusion Criteria:

* Hematologic malignancy or blood disorder requiring allogeneic HCT
* Adequate vital organ function as defined per protocol
* Karnofsky Performance Status Score (KPS) ≥ 80%
* Participants must have an available 8/8 HLA-A, -B, -C, and -DRB1 matched-related or unrelated donor

Exclusion Criteria:

* Active infection not controlled with appropriate antimicrobial therapy
* HIV, hepatitis B or C infection or known history of HIV, hepatitis B or C(all patients will be tested for HIV, hepatitis B and C as part of standard pre-transplant testing, and will be excluded from this trial if positive)
* Anti-thymocyte globulin, or cyclophosphamide administered within 14 days before or planned to receive with HCT conditioning or as part of GVHD prophylaxis in the 14 days after HCT
* Known allergic reactions to components of the study drug
* Concurrent treatment with another investigational drug
* History of thromboembolism, transient ischemic attack, stroke, myocardial infarction within 3 months preceding the transplant, or uncontrolled congestive heart failure or cardiac arrhythmias.
* Post-transplant maintenance therapies such as FLT3 inhibitor, tyrosine kinase inhibitor, JAK inhibitors etc. are not allowed if plan is to initiate such therapies <90 days post-transplant. Patient will be eligible if plan to initiate maintenance therapy is after day 90 post-transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Grade II-IV Acute Graft-versus Host Disease | 1 year post HCT
  Cumulative incidence of grade II-IV acute graft-versus-host disease (GVHD) by day 100 after hematopoietic cell transplantation (HCT). Acute GVHD severity will be determined by standard Consensus Criteria, and the cumulative incidence of grade II-IV acute GVHD will be reported through day 100 post-HCT, with relapse and death as competing risk events.

SECONDARY OUTCOMES:
Chronic Graft-versus Host Disease Through 1 Year Post HCT | 1 year post HCT
  NIH criteria defined chronic graft-versus-host disease through 1 year post-HCT. Chronic GVHD will be defined by the presence of chronic GVHD defining features, regardless of time post-HCT, in keeping with the NIH Consensus Criteria on diagnosis and staging of chronic GVHD. Individual affected organs are staged on 0-3 severity scale, and summarized for an overall global severity score. The presence of acute GVHD features defines the following subgroups: (1) late acute GVHD (sole presence of acute GVHD features after day 100 post-HCT), (2) overlap subtype of chronic GVHD (co-occurrence of chronic and acute GVHD features, and (3) classic chronic GVHD (absence of concurrent acute GVHD features).
Malignancy Relapse Post-HCT | 1 year post HCT
  Defined as hematologic relapse or any unplanned intervention (including withdrawal of immune suppression) to prevent progression of disease in patients with evidence (molecular, cytogenetic, flow cytometric, radiographic) of malignant disease after HCT.
Non-relapse Mortality | 1 year post HCT
  Defined as death in the absence of malignancy relapse post-HCT.
Overall Survival (OS) | 1 year post HCT
  Defined as time from HCT to death or censoring for last follow up.

OTHER OUTCOMES:
Glucocorticoid Exposure | 1 year post HCT
  Systemic steroid (prednisone or equivalent) dose per kg of recipient body weight will be collected at each study visit, and overall exposure determined.
Neutrophil and Platelet Engraftment | 1 year post HCT
  Stable engraftment is defined as a sustained absolute neutrophil count > 500 over 3 days, as well as a sustained platelet count of > 20 over 7 days without transfusion support. Time to engraftment is defined as time from day 0 to day of sustained engraftment per above criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Khimani, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (3):
- United States (3):
  - City of Hope Cancer Center, Duarte, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio